CLINICAL TRIAL: NCT01064843
Title: Clinical Evaluation of the Mandibular Mini-Implant Overdenture
Status: Completed | Type: Observational
Sponsor: Solventum US LLC (Industry)
Collaborators: McGill University (Other); 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: 3M ESPE CR-09-020
Record Dates: First submitted 2010-02-05; First posted 2010-02-09 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Stabilization of a Full Lower Denture; Edentulism in Lower Jaw; Lower Denture Made Within Last Few Years
Keywords: Edentulous; Edentulism; Lower denture; Mini dental implant; Imtec MDI; Denture stabilization; Case success rate of overdentures stabilized by MDI; General satisfaction of patients with this treatment; Oral health-related quality of life of these patients; Cost estimates
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 4 Imtec mini-dental implants (MDI): 4 Imtec MDI
  Interventions: Device: Imtec MDI

INTERVENTIONS:
Device: Imtec MDI — 4 Imtec MDI

SUMMARY:
Stabilization of existing full lower dentures by means of mini-dental implants (MDI). To test whether 4 mini-implants placed at the front of the lower jaw can stabilize an immediately-modified existing lower denture.

DETAILED DESCRIPTION:
To test whether the percentage of case successes of these lower dentures supported by 4 MDIs is equal to or greater than 95% at 1 year. Success is defined as a denture supported by implants that is functioning in the way it was intended.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous with last tooth extraction 2 years ago or longer.
* Patients requesting implant stabilization of existing lower conventional denture.
* Adequate space in anterior mandible for placement of 4 MDI implants.
* Able to maintain adequate oral hygiene and keep dentures clean.
* Healthy enough to have minor surgical procedures.
* Have adequate understanding of written and spoken English or French.
* Capable of providing written informed consent.

Exclusion Criteria:

* Not enough room in mandibular bone for implant height.
* Has acute or chronic symptoms of parafunctional disorders.
* History of radiotherapy to orofacial region.
* Are or have been taking bisphosphonate IV or other medications (to be evaluated by the researcher).
* Health conditions that may jeopardize treatment (to be evaluated by the researcher).
* Unable or unwilling to return for evaluations or study recalls.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Dental implant
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Success rate of mandibular overdentures supported by 4 MDIs placed in the interforaminal region in the long term. | 3 years

SECONDARY OUTCOMES:
Oral health-related quality of life and general satisfaction of patients. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Feine, DDS, MSc, HDR, Principal Investigator — Professor, Principal Investigator
Locations (1):
- Faculty of Dentistry, McGill University, Montreal, Quebec, Canada